CLINICAL TRIAL: NCT03252080
Title: Effect of Holistic Management on the Patients With Type 2 Diabetes Who Received or Did Not Receive a Short-term Intensive Education
Brief Title: Effect of Holistic Management on the Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cheng Qing-feng (Other)
Responsible Party: Sponsor-Investigator, Cheng Qing-feng, Associate professor, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HMD2017
Record Dates: First submitted 2017-08-03; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes; holistic management
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Group A) (Active Comparator): short-intensive education for one month
  Interventions: Behavioral: short-term intensive education
- Education & holistic management(Group B) (Experimental): short-intensive education for one month followed with holistic management for 6 months
  Interventions: Behavioral: short-term intensive education; Behavioral: Holistic management

INTERVENTIONS:
Behavioral: short-term intensive education — The patients of both groups are given the education classes once a week in the first month (total 4 times), 5 hours per class. The education classes are taught by a dedicated team of diabetes specialist doctors and nurses, with the contents including a basic understanding of diabetes, diabetic diet, exercise, drug treatments and blood glucose monitoring.
Behavioral: Holistic management — The specialist nurses talk individually with the patients for 10-15 min per week. The nurses ask the patients about their results of self-blood glucose monitoring, help them find the reasons of poor blood glucose control as well as answer the patient's questions.
  Arms: Education & holistic management(Group B)

SUMMARY:
Two hundreds patients with T2DM from the outpatient clinic of The First Affiliated Hospital of Chongqing Medical University will be enrolled in this study. Participating subjects will be randomly assigned into one of the 2 groups: Group A (n=100) will be placed on the short-term intensive education program alone while Group B (n=100) will be placed on the short-term intensive education as well as a holistic management for 6 months.

Diabetes education: The patients of each group will undergo designated education programs in 4 subgroups. Group A and B will be given the same education classes once a week in the first month (total 4 times), 5 hours per class. The education classes will be taught by a dedicated team of diabetes specialist doctors and nurses, with the contents including a basic understanding of diabetes, diabetic diet, exercise, drug treatments and blood glucose monitoring. At the conclusion of the education classes, the patients in Group B then will undergo a weekly telephone interview with specialist nurses for 6 months to help patients resolve self-management problems while patients in Group A will not. The specialist nurses will talk individually with the patients in Group B for 10-15 min per week. The nurses will ask the patients about their results of self-blood glucose monitoring, help them find the reasons of poor blood glucose control as well as answer the patient's questions.

Clinical examination: All subjects will complete Audit of Diabetes Dependent Quality of Life (ADDQoL) before education classes commence (baseline), at 3 months and 6 months (endpoint) after education classes to evaluate their quality of life. All patients will be examined for height, weight, blood pressure, FPG, PPG and HbA1c at baseline, 3 months after education classes and endpoint. A diabetes specialist nurse will measure the height, weight and blood pressure, and assist the subjects to fill the questionnaire. FPG and PPG will be determined by the hexokinase method, while HbA1c by high performance liquid chromatography.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM for more than 1 year,
* Age from 18 to 75 years old,
* Have fasting plasma glucose (FPG) ≥ 7.2mmol/L or 2 hours postprandial plasma glucose (2hPPG) ≥ 10.0mmol/L,
* Glycosylated hemoglobin (HbA1c) ≥ 7.0%,
* Have the ability to self-care.

Exclusion Criteria:

* Patients with severe liver or kidney dysfunction, severe heart failure, cognitive dysfunction or pregnancy will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
ADDQoL score at endpoint | 6 months
  All subjects complete Audit of Diabetes Dependent Quality of Life (ADDQoL) at endpoint to evaluate their quality of life. There are 13 items including Employment/career, Social life, Family relationships, Friends, Sex life, Sport/leisure, Travel, Future (own), Future of family, Motivation, Physical activities, Others fussing and Enjoyment of food. Each item is scored -3 to +3 (-3 = would be a great deal better if I did not have diabetes; +3 = would be a great deal worse if I did not have diabetes), yielding total between -39 to +39.

SECONDARY OUTCOMES:
Change of ADDQoL score between baseline and endpoint | 6 months
  All subjects complete Audit of Diabetes Dependent Quality of Life (ADDQoL) at baseline and endpoint to evaluate their quality of life. There are 13 items including Employment/career, Social life, Family relationships, Friends, Sex life, Sport/leisure, Travel, Future (own), Future of family, Motivation, Physical activities, Others fussing and Enjoyment of food. Each item is scored -3 to +3 (-3 = would be a great deal better if I did not have diabetes; +3 = would be a great deal worse if I did not have diabetes), yielding total between -39 to +39. The change of ADDQoL score between baseline and endpoint = the total score of ADDQoL at endpoint - the total score of ADDQoL at baseline.
FPG at endpoint | 6 months
  All patients are examined for FPG at endpoint. FPG are determined by the hexokinase method.
PPG at endpoint | 6 months
  All patients are examined for PPG at endpoint. PPG are determined by the hexokinase method.
HbA1c at endpoint | 6 months
  All patients are examined for HbA1c at endpoint. HbA1c are determined by high performance liquid chromatography.